CLINICAL TRIAL: NCT06307262
Title: European Registry of Transcatheter Repair for Tricuspid Regurgitation (EuroTR)
Brief Title: European Registry of Transcatheter Repair for Tricuspid Regurgitation
Acronym: EuroTR
Status: Recruiting | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Jörg Hausleiter, Deputy chief, LMU Klinikum
Other Study IDs: EuroTR Registry
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Tricuspid Regurgitation; Valvular Heart Disease; Heart Failure
Keywords: Tricuspid regurgitation; TEER; edge-to-edge repair
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: T-TEER — T-TEER using the PACAL or TriClip device
  Other Names: Transcatheter tricuspid valve edge-to-edge repair

SUMMARY:
To investigate clinical and survival outcomes following transcatheter tricuspid valve repair or replacement.

DETAILED DESCRIPTION:
Background and Rationale:

Tricuspid regurgitation (TR) is a major health and economic burden due to high rates of heart failure hospitalizations, morbidity and mortality. Surcial treatment of TR is associated with high procedural and in-hospital mortality. Due to prohibitive surgical risk, a significant proportion of patients historically remained untreted beyond medical therapy. Transcatheter tricuspid valve (TV) repair and replacement techniques (TTVT) now offer a new treatment perspective for these patients. The EuroTR registry aims at optimizing patient selection prior to TTVT and thus treatment quality by collecting respective data in a real-world setting.

Objectives:

To investigate clinical and survival outcome following transcatheter tricuspid valve repair or replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with one of the following transcatheter devices for TV repair or replacement: PASCAL, TriClip, TricValve, Evoque, LuX-Valve
* Age ≥ 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with one of the following transcatheter devices for TV repair or replacement (e.g. PASCAL, TriClip, TricValve, Evoque, LuX-Valve)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 5 years

SECONDARY OUTCOMES:
Technical success | 5 years
  absence of procedural mortality, successful access, delivery and retrieval of the delivery system, successful deployment and positioning, freedom from emergency surgery
Procedural Safety | 5 years
  periprocedural and in-hospital adverse events
Heart Failure Biomarker | 5 years
  NT-proBNP level
Dyspnea on exertion | 5 years
  New York Heart Association (NYHA) functional class
Functional capacity | 5 years
  6-minute walk distance (6MWD)
Right ventricular size | 5 years
  Mid-ventricular diameter of the right ventricle measured by echocardiography
Right ventricular function | 5 years
  Right ventricular fractional area change measured by echocardiography
Tricuspid regurgitation reduction | 5 years
  Tricuspid regurgitation severity measured by echocardiography
Tricuspid valve stenosis | 5 years
  Transvalvular pressure gradient measured by echocardiography
Pulmonary hypertension | 5 years
  Pulmonary artery pressure measured by echocardiography
Right heart congestion | 5 years
  Inferior vena cava dimensions measured by echocardiography
Hospitalization for heart failure | 5 years
  Date and number of heart failure hospitalizations after the index procedure

CONTACTS AND LOCATIONS:
Locations (1):
- LMU Klinikum, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masiero G, Arturi F, Ceni S, Panza A, Kresoja KP, von Stein J, Fortmeier V, Koell B, Rottbauer W, Kassar M, Goebel B, Denti P, Achouh P, Rassaf T, Barreiro-Perez M, Boekstegers P, Ruck A, Zdanyte M, Adamo M, Vincent F, Schlegel P, Rosch S, Wild MG, Besler C, Toggweiler S, Brunner S, Grapsa J, Patterson T, Thiele H, Kister T, Sticchi A, De Carlo M, Voss F, Polzin A, Popolo Rubbio A, Bedogni F, Stolte T, Nestelberger T, Benito-Gonzalez T, Sanchez-Munoz E, Konstandin MH, Van Belle E, Metra M, Geisler T, Estevez-Loureiro R, Mahabadi AA, Karam N, Maisano F, Lauten P, Praz F, Kessler M, Kalbacher D, Rudolph V, Iliadis C, Lurz P, Hausleiter J, Stolz L, Tarantini G; EuroTR Investigators. Invasive Hemodynamics and Risk Stratification in T-TEER: Moving Beyond ESC Thresholds: EuroTR Registry Insights. Circ Cardiovasc Interv. 2025 Nov 14:e015964. doi: 10.1161/CIRCINTERVENTIONS.125.015964. Online ahead of print. PMID 41235431